CLINICAL TRIAL: NCT03567096
Title: Characterization of Acute and Long Term Response to Left Ventricle Only Pacing Combined With MultiPoint Pacing and SyncAV
Brief Title: LV Only MPP With SyncAV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SJM-CIP-10231
Record Dates: First submitted 2018-05-25; First posted 2018-06-25 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Heart Failure; Left Bundle-Branch Block
Keywords: Cardiac resynchronization therapy; MultiPoint Pacing
MeSH Terms: conditions — Heart Failure; Bundle-Branch Block

STUDY DESIGN:
Intervention Model Description: Prospective, two-arm, randomized 1:1, multicenter study
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- BiV+MPP (Active Comparator): Patients randomized to the "BiV pacing with MPP and SyncAV" study arm will have CRT programming to biventricular pacing with MPP activated. RV-LV pacing delay set to 5 ms, LV1 & LV2 pacing cathodes selected as the maximal spaced electrodes (D1+P4, D2+M3, M2+P4) with pacing delay set to 5 ms and SyncAV offset programmed providing the optimum electrical resynchronization (shortest QRS duration).
  Interventions: Device: BiV pacing with MPP and SyncAV
- LV-only + MPP (Experimental): Patients randomized to the " LV only pacing with MPP and SyncAV" study arm will have CRT programming to left ventricular only pacing with MPP activated. LV1 & LV2 pacing cathodes selected as the maximal spaced electrodes (D1+P4, D2+M3, M2+P4) with pacing delay set to 5 ms and SyncAV offset programmed providing the optimum electrical resynchronization (shortest QRS duration)
  Interventions: Device: LV only pacing with MPP and SyncAV

INTERVENTIONS:
Device: BiV pacing with MPP and SyncAV — This cohort will receive Bi-Ventricular Pacing (left ventricle and right ventricle pacing) with MultiPoint Pacing of the left ventricle (two stimulation sites) and the SyncAV algorithm active.
  Arms: BiV+MPP
Device: LV only pacing with MPP and SyncAV — This cohort will receive left ventricular only pacing (no right ventricle pacing) with MultiPoint Pacing of the left ventricle (two stimulation sites) and the SyncAV algorithm active.
  Arms: LV-only + MPP

SUMMARY:
The objective of this clinical investigation is to evaluate the clinical benefits of left ventricle (LV) only pacing combined with automatic adjustment of AV timing (SyncAV) in patients receiving cardiac resynchronization therapy (CRT) after 6 months of therapy.

This clinical investigation is a prospective, two-arm, randomized 1:1, multicenter feasibility study designed to evaluate the effectiveness of LV only with multipoint pacing (MPP) and SyncAV compared to bi-ventricular pacing with MPP and SyncAV. The clinical investigation will be conducted at approximately 7 centers in Europe and Canada. Approximately 120 subjects will be enrolled in the study. No site may enroll more than 33% of the total subjects.

Data will be collected at enrollment, CRT implant procedure, hospital pre-discharge, one and 6 months post implant. Enrollment data collection will include demographics, cardiovascular history, medication, echocardiography measurements and quality of life questionnaire. CRT implant procedure data collection will include implanted system information and lead location. The electrical conduction recording procedure will include surface ECG and device IEGM recordings during various pacing configurations at implant or up to 45 days post implant. In patients who consent to invasive measurements (expected target of at least 80 patients), a hemodynamic recording procedure will include invasive hemodynamic measurements during various pacing configurations which may take place during device implant or up to 45 days post implant. Hospital pre-discharge data collection will take place within 3 days after the CRT implant, electrical conduction recordings visit or hemodynamic recordings visit and will include system information, surface ECG, and device IEGMs.

In a subset of patients from selected centers that have access to this technology (expected 20 patients), non-invasive electrical activation data will be collected with body surface mapping within 45 days of the implant procedure.

Patients will be randomized 1:1 to receive either biventricular pacing with multipoint pacing (MPP) or LV-only pacing with MPP at the one-month (± 15 days) visit. The 6-month (± 15 days) post randomization follow up visit will include surface ECG, IEGMs, echocardiographic parameters and quality of life questionnaire.

Subjects participating in this clinical investigation will follow the hospital center standard of care from implant to 6 month follow up. The expected duration of enrollment is 1.5 year. The total duration of the clinical investigation is expected to be 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with approved indication for CRT scheduled to be implanted with an MPP-enabled ABT Quadripolar CRT pacing system, de novo or upgrade from non-CRT system
* Patient must be > 18 years of age, able to provide informed consent and willing to comply with study requirements
* Documented permanent left bundle branch block (LBBB)
* Intrinsic QRS duration ≥ 150 ms
* Sinus (or atrial paced) rhythm with intact AV conduction with PR interval ≤ 250 ms

Exclusion Criteria:

* Resting heart rate > 100 bpm
* AV Block (1st degree with PR> 250 ms, 2nd or 3rd degree)
* Documented persistent atrial tachycardia or atrial fibrillation at the moment of enrollment or patients not likely to remain in sinus (or atrial paced) rhythm for the duration of the study
* Patients scheduled for AV node ablation to treat paroxysmal atrial arrhythmias
* Recent (< 3 months) myocardial infarction, ablation, electrolyte imbalance, or any condition within the last 90 days that would contraindicate for CRT programming changes in the opinion of the investigator
* Women who are pregnant or plan to become pregnant during the study course

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2018-10-09 (Actual); Primary Completion 2023-02-24 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Clinical response | up to 6 months
  Patient clinical response to LV only pacing with SyncAV optimization at six-month follow-up evaluated by the Packer clinical composite score.

SECONDARY OUTCOMES:
Left Ventricle reverse remodeling | up to 6 months
  Patient reverse remodeling response to LV only pacing at six-month follow-up defined as end-systolic volume reduction >15%.
Electrical resynchronization | intraoperative
  Acute changes in surface ECG QRS duration resulting from various CRT and SyncAV pacing configurations.

OTHER OUTCOMES:
Hemodynamic response | intraoperative
  Acute changes in LV dP/dtmax (measured with pressure wire, pressure-volume loop catheter or non-invasive system) resulting from various CRT and SyncAV pacing configurations (subset of patients consenting to invasive measurements
Left Ventricle Electrical Activation | intraoperative
  Acute changes in LV activation time resulting from various CRT and SyncAV pacing configurations (subset of patients undergoing body surface mapping).

CONTACTS AND LOCATIONS:
Overall Officials: Bernarnd Thibault, MD, Principal Investigator — Montreal Heart Institute
Locations (6):
- Montreal Heart Institute, Montreal, Canada
- CHU Rennes, Rennes, France
- Policlinico Casilino, Roma, Italy
- United Kingdom (3):
  - Queen Elizabeth Hospital, Birmingham
  - St. Bartholomew's Hospital, London
  - John Radcliffe Hospital, Oxford

IPD SHARING:
Plan to Share IPD: No
No participant data will be shared to other researchers

REFERENCES:
- [Derived] Thibault B, Waddingham P, Badie N, Mangual JO, McSpadden LC, Betts TR, Calo L, Grieco D, Leyva F, Chow A. Acute Electrical Synchronization Achieved With Dynamic Atrioventricular Delays During Biventricular and Left Ventricular MultiPoint Pacing. CJC Open. 2024 Nov 8;7(2):166-175. doi: 10.1016/j.cjco.2024.11.003. eCollection 2025 Feb. PMID 40060211